CLINICAL TRIAL: NCT06168695
Title: Impact of Anterior Dental Cross Bite Treatment on Children's Speech Performance and Their Quality of Life
Brief Title: Impact of Anterior Cross Bite Treatment on Children's Speech Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, Lecturer of Pediatric dentistry, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #R-PED-1-23-6
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cross Bite; Malocclusion; Speech; Quality of Life
Keywords: crossbite; speech; expansion screw; quality of life
MeSH Terms: conditions — Malocclusion; Speech | interventions — Quality of Life; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: prospective, single-arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anterior crossbite treatment with evaluation of speech and quality of life (Experimental): removable anterior expansion screw is used to correct anterior crossbite
  Child Perceptions Questionnaire was used to gauge how the anterior crossbite affected the children's OHRQoL.
  children were subjected to the Protocol of speech evaluation
  Interventions: Device: removable anterior expansion screw; Diagnostic Test: Speech and language evaluation; Other: Oral Health Related Quality of Life (OHRQoL) Assessment

INTERVENTIONS:
Device: removable anterior expansion screw — For the upper and lower arches, precise and profound alginate impressions were obtained and plaster study models were created. The removable appliance was constructed using acrylic resin with bilateral occlusal coverage for posterior teeth. The removable appliance was inserted in the patient's mouth and the patient was recalled after 24 hours to check the appliance fit.
  Patient was recalled every four weeks until the dental cross-bite was corrected.
Diagnostic Test: Speech and language evaluation — speech evaluation was done by a Phoniatrician and all children were subjected to the Protocol of speech evaluation before expansion screw appliance insertion and after complete correction of anterior crossbite using an articulation test, intelligibility test, and spectrographic analysis.
  * Articulation test: Five speech sounds were chosen to be studied /s/, /s /, /z/, /z/, /∫ /. The consonants were tested in the initial, medial, and final word positions.
  * Speech intelligibility test : The general intelligibility score was calculated using Speech intelligibility in context: 5 -point scale:
  * Spectrographic analysis: Using the computerized speech lab, the child was seated in an upright position & allowed to talk freely & repeated syllables were said to him/her.
Other: Oral Health Related Quality of Life (OHRQoL) Assessment — The Child Perceptions Questionnaire (CPQ 8-10) in Brazilian version was used to gauge how the anterior cross bite affected the children's OHRQoL. It has twenty-five items total, broken down into four health domains (subscales): five questions each about oral symptoms (OS), five questions about functional limitations (FL), five questions about emotional wellbeing (EW), and ten questions about social well-being (SW). The responses never (0), once/twice (1), occasionally (2), often (3), and every day/almost every day (4) are provided for each question on an ordinal scale. The sum of the scores for all questions is used to calculate the scores for each subscale. The CPQ 8-10 was used to assess the OHRQoL before appliance insertion and after complete correction of anterior crossbite.

SUMMARY:
The goal of this prospective, single-arm clinical trial is to evaluate the speech performance of children with anterior dental crossbite before and after correction. Also, to assess the impact of early interceptive orthodontic treatment in the mixed dentition stage to correct the anterior dental crossbite on the quality of life of children.

Fifty children of both sexes aged from 8 to 10 years were enrolled and evaluated using the study's inclusion & exclusion criteria. before beginning interceptive orthodontic treatment, each child underwent full mouth treatment. then, using a removable anterior expansion screw along with posterior bite planes to treat the anterior crossbite. All children were subjected to the Protocol of speech evaluation before appliance insertion and after complete correction of anterior crossbite. Also, the Child Perceptions Questionnaire (CPQ 8-10) in the Brazilian version was used to gauge how the anterior crossbite affected the children's oral health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* healthy cooperative children aged 8-10 years
* have at least one or more maxillary permanent incisors in a crossbite relationship
* fully erupted four first permanent molars
* Angle Class I molar relationship and Class I skeletal relationship
* the mother language of all the subjects was Arabic.

Exclusion Criteria:

* Children with systemic illness or previous history of speech therapy
* children who are ill-habituated or unable to follow up
* children with previous orthodontic treatment
* uncooperative children
* Anterior skeletal or functional crossbite
* presence of sucking habits

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-02-04 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
normal anterior occlusion, no anterior crossbite, normal measured Overjet and Overbite | 3 months
  Normal occlusion is measured as:
  no anterior crossbite Overbite 1 mm to 4 mm Overjet 1mm to 4 mm

SECONDARY OUTCOMES:
child compliance, oral health-related quality of life questionnaire | 3 months
  The earlier tested questionnaire is used to compare child compliance before and after anterior crossbite correction
Measured degree of speech improvement | 3 months
  The pre-treatment assessed speech sounds are compared with the post-treatment assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Littlewood SJ, Tait AG, Mandall NA, Lewis DH. The role of removable appliances in contemporary orthodontics. Br Dent J. 2001 Sep 22;191(6):304-6, 309-10. doi: 10.1038/sj.bdj.4801170. PMID 11587502
- [Background] Assaf DDC, Knorst JK, Busanello-Stella AR, Ferrazzo VA, Berwig LC, Ardenghi TM, Marquezan M. Association between malocclusion, tongue position and speech distortion in mixed-dentition schoolchildren: an epidemiological study. J Appl Oral Sci. 2021 Aug 16;29:e20201005. doi: 10.1590/1678-7757-2020-1005. eCollection 2021. PMID 34406316
- [Background] Jokovic A, Locker D, Stephens M, Kenny D, Tompson B, Guyatt G. Validity and reliability of a questionnaire for measuring child oral-health-related quality of life. J Dent Res. 2002 Jul;81(7):459-63. doi: 10.1177/154405910208100705. PMID 12161456